CLINICAL TRIAL: NCT06819267
Title: Horizontal Versus Vertical Plyometric Exercises On Agility, Speed And Power Among Rugby Players
Brief Title: Effects Of Horizontal Versus Vertical Plyometric Exercises On Agility, Speed And Power Among Rugby Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0419
Record Dates: First submitted 2025-01-10; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horizontal Plyometric Group (Experimental)
  Interventions: Other: Horizontal Plyometric Group
- Vertical Plyometric Group (Experimental)
  Interventions: Other: Vertical Plyometric Group

INTERVENTIONS:
Other: Horizontal Plyometric Group — Group A
  * Duration: A 30-minute treatment session for four weeks.
  * Frequency: Two to three sessions per week.
  * Warm-up: 5 minutes following the FITT principle (Frequency, Intensity, Time, Type).
  * Warm-up Components:
  * 5 minutes of moderate to high-intensity cardiovascular warm-up.
  * Exercise Components (30 minutes per session):
  * Horizontal ankle jumps| Long jumps | Diagonal obstacle jumps
  * Intensity: Moderate to high.
  Arms: Horizontal Plyometric Group
Other: Vertical Plyometric Group — Group B
  * Duration: A 30-minute treatment session for four weeks.
  * Frequency: Two to three sessions per week.
  * Warm-up: 5 minutes following the FITT principle (Frequency, Intensity, Time, Type).
  * Warm-up Components:
  * 5 minutes of moderate to high-intensity cardiovascular warm-up.
  * Exercise Components (30 minutes per session):
  * Vertical ankle jumps
  * Counter movement jump
  * Front obstacle jumps
  Arms: Vertical Plyometric Group

SUMMARY:
Participating in rugby demands specialized skills that encompass explosive movements and diverse muscle actions at varying speeds. Attributes like strength, speed, jumping capability, and agility play crucial roles in executing fundamental rugby skills, including sudden changes of direction, acceleration, and deceleration. Previous research has substantiated the positive impacts of plyometric training in young athletes during the in-season period, indicating the significance of targeted training during this timeframe for sustaining or amplifying explosiveness. Moreover, there is supporting evidence that integrating plyometric training into a traditional rugby training regimen yields favorable outcomes, specifically benefiting speed, vertical jumping performance, and agility. To determine the effects of horizontal versus vertical plyometric exercises on agility, speed, and power among rugby players.

This randomized clinical trial, to be carried out in DHA Rugby Stadium, Lahore, will enlist participants aged 18 to 28, encompassing both males and females, with a minimum of 1 year of rugby experience. The study aims to investigate the impact of horizontal and vertical plyometric exercises on agility, speed, and power in rugby players. Participants will be randomly assigned to Group A, receiving horizontal plyometric exercises, or Group B, receiving vertical plyometric exercises. Evaluation will involve the Hexagon test for agility, the 20m Sprint test for speed, and Vertical jump assessment for power. The results aim to contribute substantiated insights into the pre and post effects of these plyometric exercises on rugby players. Data analysis will be conducted using IBM SPSS Statistics 26

DETAILED DESCRIPTION:
To determine effects of horizontal versus vertical plyometric exercises on agility, speed, and power among rugby players.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-28
* Both genders
* Rugby Players (playing 2 to 3 days per week)

Exclusion Criteria:

* Players with any previous injury
* Any congenital disorder
* Not playing for more than 6 months
* Symptoms of coronary artery and pulmonary disease

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
A Haxagon test for agility | 4 weeks
  The Hexagon Agility Test is a physical assessment that evaluates an individual's agility, quickness, and ability to change direction rapidly. It typically involves a hexagon-shaped pattern marked on the ground. The participant stands at the center of the hexagon, and on a signal, moves quickly to touch each of the six corners and return to the center.
A Vertical Jump test | 4 weeks
  The Vertical Jump test assesses an individual's lower body power by measuring how high they can jump vertically. The participant stands next to a wall or a vertical measuring device and jumps as high as possible, reaching upward with their arm closest to the wall to mark the highest point touched.
A 20m Sprint Test | 4 weeks
  The 20m Sprint Test for speed is a fitness assessment that measures an individual's acceleration and maximal sprinting speed over a distance of 20 meters. The participant starts from a stationary position and sprints as fast as possible to cover the designated distance

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul memon MS, MS Sports, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No